CLINICAL TRIAL: NCT04748380
Title: Shared Decision-making and Colorectal Cancer Screening Behaviors Among Older Adults With Low Health Literacy
Brief Title: Shared Decision-making and Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Tamara J. Cadet, PhD, LICSW, MPH, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UPCC 11223; 850357 (Other: University of Pennsylvania Institutional Review Board)
Record Dates: First submitted 2021-01-22; First posted 2021-02-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
Keywords: decision aid; screening; older adults; low health literacy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Stratifying by sex, 30 participants will be randomized to receive the CRC DA pamphlet and 30 will be randomized to receive the home safety information at the visit in case they cancel their appointment and reschedule.
Who Masked: Participant
Masking Description: Stratifying by sex, 30 participants will be randomized to receive the CRC DA pamphlet and 30 will be randomized to receive the home safety information at the visit in case they cancel their appointment and reschedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRC DA (Experimental): Stratifying by sex, 30 participants will be randomized to receive the CRC DA pamphlet.
  Interventions: Other: CRC decision aid pamphlet
- Home Safety Pamphlet (Other): Stratifying by sex, 30 will be randomized to receive the home safety information at the visit.
  Interventions: Other: Home Safety Pamphlet

INTERVENTIONS:
Other: CRC decision aid pamphlet — A newly developed 8-10 page decision aid pamphlet that discusses:1. Information on CRC; 2. Information about risk and benefits including the 10-year lag-time to benefitting from CRC screening; 3. Information to help patients evaluate CRC screening options (colonoscopy or stool testing); 4. Possible outcomes relevant to LE and health status. In addition, there will be a values clarification exercise
  Arms: CRC DA
Other: Home Safety Pamphlet — The home safety information pamphlet is a 2-page fact sheet on home safety tips for older adults, and was designed by the AGS Health in Aging Foundation. It includes information in seven areas to help older adults stay safe in their homes. Areas include but are not limited to fall prevention and safety proofing homes. It has been used successfully in prior studies of DAs as a control intervention
  Arms: Home Safety Pamphlet

SUMMARY:
Conduct a feasibility pilot RCT of a newly developed colorectal cancer screening (CRC) decision aid (DA) including 66 LHL adults 76-85 years recruited from community health centers. Hypotheses: Patients in the intervention group will be more likely to change their intentions to be screened with fewer patients with <10 year LE and/or those with >10 year LE and no risk factors intending to be screened and more with >10 year LE and risk factors for CRC and/or those who have never been screened intending to be screened (primary outcome). The secondary outcomes are that the patients in the intervention group will have 1. increased knowledge of CRC screening options and the benefits and risks of these options; 2. increased SDM engagement; and 3. find the DA acceptable. Investigators also anticipate that at least 50% of eligible participants will choose to participate in the study.

DETAILED DESCRIPTION:
Investigators will recruit and survey 66 adults (to reach a goal of 60 with complete data), 75-85 years with low health literacy LHL (30 per arm) over 24 months to learn the effects of the newly developed CRC DA pamphlet on older adult's screening intentions, knowledge of options and the benefits and harms, and SDM from community health centers. Investigators collect baseline data over the phone prior to the visit. Patients who are eligible and willing to participate will come to a regularly scheduled visit with their primary care physician (PCP) early to answer the pretest questions. Stratifying by sex, 30 participants will be randomized to receive the CRC DA pamphlet and 30 will be randomized to receive the home safety information at the visit in case they cancel their appointment and reschedule. The home safety information is 2 pages, and was designed by AGS Health in Aging Foundation. It has been used successfully in prior studies of DAs as a control intervention. Investigators chose this pamphlet for the control arm because it is written at <7th grade reading level and reading about home safety should not affect screening decisions. Providing the control group the home safety pamphlet to read reduces response bias since it helps keep participants blinded to the intervention of interest and compensates for the time and attention required by the intervention group to read the DA. At the visit, participants will review the DA or the home safety pamphlet. The revised CRC DA pamphlet is expected to take 5-10 minutes to read as well as the home safety pamphlet. After completing the pre-survey questionnaire before the visit the patient will have their PCP visit. The post-test will be asked after the PCP visit in person or over the phone (depending on the participant's preference, access to a phone, and ability to stay after their appointment for enough time to complete the post-visit questionnaire). Investigators will conduct a chart review at 6 months to see if a CRC screening discussion occurred and the outcome (i.e., qualitative trends in use of CRC screening). Investigators will also call each patient at 6 months to ask about their CRC screening intentions.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 75 and 85 years
* Must be low health literacy (LHL), determined by participants' response to the validated LHL question, "How confident are you filling out medical forms by yourself?" with a response of, "somewhat to not at all confident."39-43
* Have an educational level at community college or less

Exclusion Criteria:

* Patients who do not have the capacity to participate
* Patients with dementia
* Patients with a history of invasive/non-invasive colorectal cancer.
* Patients older than 85 years since guidelines recommend against CRC screening in this age range.

Ages: 75 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Change in CRC Screening Intentions | Baseline, pre-intervention to immediately after the intervention
  Number of participants who indicate their intentions to be screened or not be screened for CRC, Change from baseline to immediately after the intervention

SECONDARY OUTCOMES:
Change in Knowledge | Baseline, pre-intervention to immediately after the intervention
  Number of participants who correctly answer 15 true/false knowledge questions developed the investigators, about the harms and benefits of CRC screening, Change from baseline to immediately after the intervention
Perceptions of Shared Decision-making Role | immediately after the intervention
  Number of participants who answer the question that participants want to make a CRC screening decision with their physician, from 5 decision-making role questions developed the investigators
Perceptions of the Length of the Decision Aid | immediately after the intervention
  Number of participants who indicate the decision aid is the right length, from a likert-scale question
Perceptions of the Clarity of the Decision Aid | immediately after the intervention
  Number of participants who indicate the decision aid is clear in the information presented, from a likert-scale question
Perceptions of the Balance of the Decision Aid | immediately after the intervention
  Number of participants who indicate the decision aid present information that is not slanted towards CRC screening or slanted away from CRC screening, from a likert-scale question
Feelings of anxiety when reading the decision aid | immediately after the intervention
  Number of participants who felt anxious after reading the decision aid, from a likert-scale question
Feelings of usefulness of the decision aid | immediately after the intervention
  Number of participants who indicate recommending the decision aid to a friend, from a likert-scale question

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available to other researchers.